CLINICAL TRIAL: NCT03928886
Title: Discomfort Assessment of Senographe Pristina Patient-assisted Versus Standard Compression Mode in Asymptomatic Adult Women Undergoing Screening Full-filled Digital Mammography and Quality Evaluation of Screening Mammograms
Brief Title: Discomfort Assessment of Senographe Pristina Patient-assisted Versus Standard Compression Mode and Quality Assessment of Screening Mammograms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Parc de Salut Mar (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Screening
Other Study IDs: 2017-7631
Record Dates: First submitted 2019-04-16; First posted 2019-04-26 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Mammography Related Discomfort
Keywords: discomfort; patient-assisted compression; breast cancer; screening; mammography; Senographe Pristina
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Each subject will undergo her regularly scheduled full-field digital mammography imaging exam per standard practices at the investigational site. Study-related compressions will consist of the first and second CC and MLO compressions performed on each breast during each subject's exam. Both the laterality (right/left breast) to which compression modes are assigned and the mode of compression to start with will be randomized across all subjects. Hence, approximately one quarter of women will use patient-assisted compression as first option on the right breast, another quarter will use patient-assisted compression as first option on the left breast, a third quarter will use standard compression as first option on the right breast and the last quarter will use standard compression as first option on the left breast. The randomization schedule will be generated by Epidemiology and Evaluation Department of the Hospital and provided to the study staff prior to start of enrollment.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Senographe Pristina patient-assisted compression model (Experimental): Senographe Pristina is a commercial mammography medical device consisting of the Senographe Pristina FFDM system (2D) and Senographe Pristina DBT option (3D). Senographe Pristina includes the hardware and software components required for multi-modality functioning and is designed to improve patient experience, patient throughput, and radiographer experience. The system offers two compression modes - standard mode and the optional patient-assisted compression. The patient-assisted compression feature enables the patient to personally refine breast compression using a hand-held remote control after the compression has been initiated by the operator, which is required to ensure proper breast positioning.
  Interventions: Device: bilateral two-view (CC and MLO) FFDM (full field digital mammography) using patient-assisted compression mode
- Senographe Pristina standard compression mode (usual care) (Active Comparator): Senographe Pristina standard mode
  Interventions: Device: bilateral two-view (CC and MLO) FFDM (full field digital mammography) using standard compression mode

INTERVENTIONS:
Device: bilateral two-view (CC and MLO) FFDM (full field digital mammography) using patient-assisted compression mode — Patient-assisted mode of Senographe Pristina (a commercial mammography medical device consisting of the Senographe Pristina FFDM system -2D- and Senographe Pristina DBT option -3D-) for FFDM imaging procedure. The patient-assisted compression feature enables the patient to personally refine breast compression using a hand-held remote control after the compression has been initiated by the operator, which is required to ensure proper breast positioning.
  Arms: Senographe Pristina patient-assisted compression model
Device: bilateral two-view (CC and MLO) FFDM (full field digital mammography) using standard compression mode — Standard compression mode of Senographe Pristina (a commercial mammography medical device consisting of the Senographe Pristina FFDM system -2D- and Senographe Pristina DBT option -3D-) for FFDM imaging procedure.
  Study-related compressions will consist of the first and second CC and MLO compressions performed on each breast during each subject's exam.
  Arms: Senographe Pristina standard compression mode (usual care)

SUMMARY:
Senographe Pristina is a new mammography system (hardware and software) designed to improve patient experience, patient throughput, and radiographer experience while maintaining the imaging capabilities and image quality of full-field digital mammography (FFDM) and digital breast tomosynthesis (DBT) breast imaging. The purpose of this study is to assess patient experience as it relates to discomfort when patient-assisted compression is compared against the standard compression mode of Senographe Pristina in asymptomatic adult women undergoing screening FFDM mammography.

The technical/clinical quality assessment of mammograms is essential to ensure that high quality images are consistently used in a breast cancer screening program. Advances in mammography equipment may improve the image quality. Therefore, the investigators hypothesize that the introduction of Senographe Pristina may have an effect on the technical/clinical quality of screening mammograms.

DETAILED DESCRIPTION:
Leading authorities on breast cancer recommend regular screening mammography for women aged 40 years and older as a means of early detection for breast cancer, which can lead to increased survival rates and more treatment options. Numerous randomized trials have demonstrated that regular mammographic screening reduces breast cancer mortality, with more than 40% reduction in breast cancer deaths. Amidst the success of screening mammography, clinicians struggle to maintain patient participation in regular screening programs. Notably, a systematic review by Whelehan, et al. concluded that pain experienced during screening mammography (e.g. compression pain) contributed to reduced rates of repeat participation in regular screening programs.

Adequate breast compression during mammography creates uniform thickness and flattens tissues, which is necessary to obtain sufficient image quality and reduce radiation dose. Various methods are being investigated to maintain sufficient compression while reducing pain associated with mammography. Specifically, studies have shown that a personalized approach to compression can significantly reduce pain intensity and discomfort experienced by patients while maintaining diagnostic image quality.

Patient-controlled compression allows the patient to control the amount of compression force during mammography and is a personalized approach that has demonstrated successful pain reduction in mammography. GE Healthcare's Senographe Pristina, an innovative mammography platform that provides both two-dimensional (2D) and three-dimensional (3D) imaging capabilities, offers standard and patient-controlled compression modes. The study described herein is being conducted to compare discomfort experienced by asymptomatic women undergoing full-field digital (FFDM) 2D screening mammography with standard and patient-controlled compression modes of Senographe Pristina. Results from this study may be used to support future regulatory submissions.

The population of this study will consist of adult asymptomatic women presenting for screening FFDM. Eligible patients will be enrolled and will undergo bilateral two-view (CC and MLO) imaging with Senographe Pristina.

Each subject will use both standard and patient-assisted compression modes, with one mode randomly assigned to the right breast and the other mode assigned to the left breast. Immediately following image acquisition (i.e. during decompression), subjects will be asked to rate their level of discomfort using a validated 11-point pain rating scale (numeric rating scale). Additional data collected from each subject will include demographic and clinical history information, breast thickness, radiation dose, compression force, and overall patient experience feedback.

Pain scores will be summarized with descriptive statistics and other endpoint data will be analyzed using general statistical methods. Pain results will be compared according to compression mode and multivariate analysis will be performed to assess the potential effect of other variables. The technical/clinical quality assessment of mammograms is essential to ensure that high quality images are consistently used in a breast cancer screening program. Poor image quality may lead to missed diagnoses and compromised detection of breast cancers. In this sense, it has been reported that high image quality leads to higher detection rates and fewer interval cancers.

In order to assess the technical/clinical quality of screening mammograms, the PGMI (perfect, good, moderately good, and inadequate) system will be used. With this system the investigators routinely evaluate the technical/clinical quality of screening mammograms in our center. A random sample of 500 women with two (2) Medio Lateral Oblique (MLO) and two (2) Cranial Caudal (CC) views produced with Senographe Pristina (291 with patient-assisted compression and 291 with standard compression mode) will be assessed by three highly trained radiologists. Technical/clinical image quality will be compared according to compression mode and multivariate analysis will be performed to assess the potential effect of other variables. Additionally, the investigators will compare the technical/clinical image quality of mammograms produced by Senographe Pristina with the image quality observed in the previous routine evaluations performed in our center.

ELIGIBILITY:
Inclusion Criteria:

* Women participating in their subsequent round in the breast cancer screening program
* Asymptomatic women scheduled for full-field digital screening mammography
* Have left and right breasts
* Have breast sizes compatible with the dimensions of a 24x29 cm image detector without anatomical cut-off
* Are able to provide subjective pain scores, per verbal self-report
* Are documented as non-pregnant based on the investigator's medical judgment and in consideration of local clinical practice standards for evidence of non-pregnancy
* Are able and willing to comply with study procedures
* Are able and willing to provide written informed consent to participate

Exclusion Criteria:

* Have been previously included in this study or are participating in another study expected to interfere with study procedures or outcomes;
* Have undergone diagnostic or surgical intervention(s) or procedure(s) on either breast, including breast biopsy, lumpectomy or mastectomy, or reconstruction;
* Are currently undergoing radiotherapy or chemotherapy, or have a history of prior radiotherapy treatment on either breast;
* Are currently lactating
* Have breast implants.

Ages: 50 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Patient discomfort using an 11-point numeric pain rating scale | Immediately following full-field digital mammography breast imaging
  Subject-provided pain scores using an 11-point numeric rating scale (NRS) of patient-assisted compression and standard compression will be used as a measure of discomfort. A total of six (6) pain scores will be obtained from each subject, consisting of two (2) baseline pain scores (right/left breast) collected previous to the image acquisition, two (2) patient-assisted compression scores (CC and MLO) and two (2) standard compression scores (CC and MLO). Immediately following image acquisition (i.e. during decompression of the breast), study staff will ask the subject to provide a verbal score, indicating her level of pain for the given compression. A validated 11-point NRS will be used for each assessment, where a score of 0 will indicate no pain and 10 will indicate the worst pain. Pain scores will be documented on Case Report Form (CRFs) by the study staff

SECONDARY OUTCOMES:
Technical/Clinical quality of mammogram using the PGMI system | Immediately following radiologists analysis
  Two highly trained radiologists will independently assess the quality of the images according to the PGMI system (Perfect, Good, Moderate, Inadequate). In case of disagreement, a third radiologist will assess the quality and a final score will reach by majority. All participating radiologists will be blind to the compression status. Items taken into account for the PGMI are: (i) For CC view: Nipple not in profile, skin folds, images not symmetrical, medial border of the breast not seen, axillary tail of the breast insufficiently seen, inadequate compression/blur, artefacts and incorrect annotation/labeling.(ii) For MLO view: insufficient inframammary angle, nipple not in profile, images not symmetrical, pectoralis major muscle not to nipple level, pectoralis major muscle not at appropriate angle, inadequate compression/blur, and artefacts. Technical/Clinical quality of mammogram using the PGMI system will be documented on CRF by the study staff
Average glandular dose in mGy | Immediately following full-field digital mammography breast imaging
  Average glandular dose is provided systematically by the mammography device following image acquisition. Results are expressed in miligray (mGy). Average glandular dose will be documented on CRF by the study staff
Breast thickness in mm | Immediately following full-field digital mammography breast imaging
  Breast thickness is provided systematically by the mammography device following image acquisition. Results are expressed in milimeters (mm). Breast thickness will be documented on CRF by the study staff
Compression force in daN | Immediately following full-field digital mammography breast imaging
  Compression force is provided systematically by the mammography device following image acquisition. Results are expressed in decanewton (daN). Compression force will be documented on CRF by the study staff.

OTHER OUTCOMES:
Patient experience feedback: Patient preference about patient-assisted compression over standard compression using a 5-point Likert scale | Immediately following full-field digital mammography breast imaging
  Study staff will provide an online questionnaire to each of the subjects when their imaging exams are completed. Subjects will complete the questionnaires while still at the site, and a member of the study staff will be available to address any questions.
  The questionnaire will consist of four (4) items, structured as statements and answered using a 5-point Likert scale: 1. Strongly agree, 2. Agree; 3. Neither agree nor disagree; 4. Disagree; 5. Strongly disagree.
  This item's statement is as follows: I preferred the patient-assisted compression exam over the standard compression exam
Patient experience feedback: Patient-assisted compression discomfort as compared to standard compression using a 5-point Likert scale | Immediately following full-field digital mammography breast imaging
  Study staff will provide an online questionnaire to each of the subjects when their imaging exams are completed. Subjects will complete the questionnaires while still at the site, and a member of the study staff will be available to address any questions.
  The questionnaire will consist of four (4) items, structured as statements and answered using a 5-point Likert scale: 1. Strongly agree, 2. Agree; 3. Neither agree nor disagree; 4. Disagree; 5. Strongly disagree.
  This item's statement is as follows: The patient-assisted compression screening exam caused less discomfort than the standard compression exam
Patient experience feedback: Expected comfortability in next screening if patient-assisted compression were available using a 5-point Likert scale | Immediately following full-field digital mammography breast imaging
  Study staff will provide an online questionnaire to each of the subjects when their imaging exams are completed. Subjects will complete the questionnaires while still at the site, and a member of the study staff will be available to address any questions.
  The questionnaire will consist of four (4) items, structured as statements and answered using a 5-point Likert scale: 1. Strongly agree, 2. Agree; 3. Neither agree nor disagree; 4. Disagree; 5. Strongly disagree.
  This item's statement is as follows: I would feel more comfortable going to my next breast screening exam if patient-assisted compression were available
Patient experience feedback: Patient-assisted compression satisfaction, expressed as the level of agreement to recommend it to friends and family using a 5-point Likert scale | Immediately following full-field digital mammography breast imaging
  Study staff will provide an online questionnaire to each of the subjects when their imaging exams are completed. Subjects will complete the questionnaires while still at the site, and a member of the study staff will be available to address any questions.
  The questionnaire will consist of four (4) items, structured as statements and answered using a 5-point Likert scale: 1. Strongly agree, 2. Agree; 3. Neither agree nor disagree; 4. Disagree; 5. Strongly disagree.
  This item's statement is as follows: I would recommend a patient-assisted compression exam to my friends and family

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Alcántara, MD, Principal Investigator — RAlcantara@parcdesalutmar.cat
Locations (1):
- Hospital del Mar - Parc de Salut Mar, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Cancer Society, "Breast Cancer Facts & Figures 2015-2016," United States, 2015.
- [Background] Nelson HD, Tyne K, Naik A, Bougatsos C, Chan BK, Humphrey L; U.S. Preventive Services Task Force. Screening for breast cancer: an update for the U.S. Preventive Services Task Force. Ann Intern Med. 2009 Nov 17;151(10):727-37, W237-42. doi: 10.7326/0003-4819-151-10-200911170-00009. PMID 19920273
- [Background] Shapiro S, Strax P, Venet L. Periodic breast cancer screening in reducing mortality from breast cancer. JAMA. 1971 Mar 15;215(11):1777-85. No abstract available. PMID 5107709
- [Background] Hendrick RE, Smith RA, Rutledge JH 3rd, Smart CR. Benefit of screening mammography in women aged 40-49: a new meta-analysis of randomized controlled trials. J Natl Cancer Inst Monogr. 1997;(22):87-92. doi: 10.1093/jncimono/1997.22.87. PMID 9709282
- [Background] Thurfjell EL, Lindgren JA. Breast cancer survival rates with mammographic screening: similar favorable survival rates for women younger and those older than 50 years. Radiology. 1996 Nov;201(2):421-6. doi: 10.1148/radiology.201.2.8888234.
- [Background] Tabar L, Vitak B, Chen HH, Yen MF, Duffy SW, Smith RA. Beyond randomized controlled trials: organized mammographic screening substantially reduces breast carcinoma mortality. Cancer. 2001 May 1;91(9):1724-31. doi: 10.1002/1097-0142(20010501)91:93.0.co;2-v. PMID 11335897
- [Background] Swedish Organised Service Screening Evaluation Group. Reduction in breast cancer mortality from organized service screening with mammography: 1. Further confirmation with extended data. Cancer Epidemiol Biomarkers Prev. 2006 Jan;15(1):45-51. doi: 10.1158/1055-9965.EPI-05-0349. PMID 16434585
- [Background] Coldman A, Phillips N, Wilson C, Decker K, Chiarelli AM, Brisson J, Zhang B, Payne J, Doyle G, Ahmad R. Pan-Canadian study of mammography screening and mortality from breast cancer. J Natl Cancer Inst. 2014 Oct 1;106(11):dju261. doi: 10.1093/jnci/dju261. Print 2014 Nov. PMID 25274578
- [Background] Hofvind S, Ursin G, Tretli S, Sebuodegard S, Moller B. Breast cancer mortality in participants of the Norwegian Breast Cancer Screening Program. Cancer. 2013 Sep 1;119(17):3106-12. doi: 10.1002/cncr.28174. Epub 2013 May 29. PMID 23720226
- [Background] Whelehan P, Evans A, Wells M, Macgillivray S. The effect of mammography pain on repeat participation in breast cancer screening: a systematic review. Breast. 2013 Aug;22(4):389-94. doi: 10.1016/j.breast.2013.03.003. Epub 2013 Mar 28. PMID 23541681
- [Background] Dullum JR, Lewis EC, Mayer JA. Rates and correlates of discomfort associated with mammography. Radiology. 2000 Feb;214(2):547-52. doi: 10.1148/radiology.214.2.r00fe23547. PMID 10671609
- [Background] Gupta R, Nayak M, Khoursheed M, Roy S, Behbehani AI. Pain during mammography: impact of breast pathologies and demographic factors. Med Princ Pract. 2003 Jul-Sep;12(3):180-3. doi: 10.1159/000070756. PMID 12766337
- [Background] Poulos A, Rickard M. Compression in mammography and the perception of discomfort. Australas Radiol. 1997 Aug;41(3):247-52. doi: 10.1111/j.1440-1673.1997.tb00668.x. PMID 9293675
- [Background] Kornguth PJ, Rimer BK, Conaway MR, Sullivan DC, Catoe KE, Stout AL, Brackett JS. Impact of patient-controlled compression on the mammography experience. Radiology. 1993 Jan;186(1):99-102. doi: 10.1148/radiology.186.1.8416595.
- [Background] de Groot JE, Broeders MJ, Branderhorst W, den Heeten GJ, Grimbergen CA. Mammographic compression after breast conserving therapy: controlling pressure instead of force. Med Phys. 2014 Feb;41(2):023501. doi: 10.1118/1.4862512. PMID 24506652
- [Background] de Groot JE, Branderhorst W, Grimbergen CA, den Heeten GJ, Broeders MJM. Towards personalized compression in mammography: a comparison study between pressure- and force-standardization. Eur J Radiol. 2015 Mar;84(3):384-391. doi: 10.1016/j.ejrad.2014.12.005. Epub 2014 Dec 13. PMID 25554008
- [Background] S. Hofvind, "Quality assurance of mammograms in the Norwegian Breast Cancer Screening Program.," European Journal of Radiology, 2009.
- [Background] Taplin SH, Rutter CM, Finder C, Mandelson MT, Houn F, White E. Screening mammography: clinical image quality and the risk of interval breast cancer. AJR Am J Roentgenol. 2002 Apr;178(4):797-803. doi: 10.2214/ajr.178.4.1780797. PMID 11906848
- [Background] Williamson A, Hoggart B. Pain: a review of three commonly used pain rating scales. J Clin Nurs. 2005 Aug;14(7):798-804. doi: 10.1111/j.1365-2702.2005.01121.x. PMID 16000093
- [Background] Li Y, Poulos A, McLean D, Rickard M. A review of methods of clinical image quality evaluation in mammography. Eur J Radiol. 2010 Jun;74(3):e122-31. doi: 10.1016/j.ejrad.2009.04.069. Epub 2009 May 30. PMID 19482454
- [Background] M. Boyce, "Comparing the use and interpretation of PGMI scoring to assess the technical quality of screening mammograms in the UK and Norway," Radiography, 2015.